CLINICAL TRIAL: NCT05491499
Title: Assessing the Impact of Exercise Based Intensive Interdisciplinary Pain Treatment (IIPT) on Endogenous Pain Modulation in Youth With Chronic Pain Syndromes
Status: Completed | Type: Observational
Sponsor: Boston Children's Hospital (Other)
Collaborators: APTA Pediatrics (Unknown)
Responsible Party: Principal Investigator, Julie Shulman, Physical Therapy Scientist, Boston Children's Hospital
Other Study IDs: P00043035
Record Dates: First submitted 2022-08-04; First posted 2022-08-08 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pain Syndrome; Fibromyalgia; Chronic Headache Disorder; Functional Abdominal Pain Syndrome; Complex Regional Pain Syndromes
MeSH Terms: conditions — Fibromyalgia; Complex Regional Pain Syndromes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Youth with Chronic pain: We will recruit 38 youth with primary and secondary chronic pain syndromes[29; 31] ages 10-17 years who are admitted to the Mayo Family Pediatric Pain Rehabilitation Center at Boston Children's Hospital. This longitudinal cohort study will examine responses to the OA and Fitkids Treadmill tests at 2 timepoints: 1) within 5 days of IIPT admission and 2) within 1 week of IIPT discharge. Twelve participants will complete a 3rd visit within 5 days of the first study visit to examine OA test-retest reliability.

SUMMARY:
This work will answer two critical questions: 1) Does intensive interdisciplinary pain treatment (IIPT) involving aerobic exercise help normalize pain processing in youth with chronic pain syndromes and 2) Are aerobic fitness levels and the ability to modulate pain inter-related?

Currently, medications are ineffective for improving pain and disability in youth with chronic pain syndromes and identifying non-pharmacologic treatments, such as IIPT, that help strengthen the nervous system's ability to modulate or turn pain signals down will improve outcomes and quality of life for youth suffering from chronic pain. This study will help determine whether exercise based IIPT leads to physiologic improvements in how pain is processed, specifically if youth with chronic pain can better turn pain down during the offset analgesia test after an exercise based IIPT treatment, and also help elucidate the link between a child's aerobic fitness and their ability to modulate pain.

DETAILED DESCRIPTION:
1. Study Design: We will recruit 38 youth with primary and secondary chronic pain syndromes[29; 31] ages 10-17 years who are admitted to the Mayo Family Pediatric Pain Rehabilitation Center (PPRC) at Boston Children's Hospital. This longitudinal cohort study will examine responses to the OA and Fitkids Treadmill tests at 2 timepoints: 1) within 5 days of IIPT admission and 2) within 1 week of IIPT discharge. Twelve participants will complete a 3rd visit within 5 days of the first study visit to examine OA test-retest reliability.
2. Description of Study Treatments or Exposures/Predictors:

Thermal testing: A computer-controlled temperature paradigm is programmed to deliver each stimulus using the Medoc Thermosensory Analyzer (TSA)-II device (Medoc Ltd. Advanced Medical Systems, Ramat Yishai, Israel). The device operates by a microcomputer-driven 3 cm x 3 cm (9 cm2) Peltier contact thermode secured to the skin by a Velcro band without stretch. Testing is conducted on the non-dominant forearm using 4 locations to minimize skin sensitivity. Participants are blinded to the type of test being performed and expected response patterns.

Assessment of Pain Intensity: During all tests participants rate heat pain intensity continuously in real time using a linear electronic visual analogue scale (eVAS). Participants use their dominant hand to operate a knob on a horizontal sliding eVAS scale (0-100 mm) with the following two anchors: the left defined as "no heat pain sensation" (0 mm) and the right as "most intense heat pain sensation imaginable" (100 mm). Participants are instructed to move the knob on the scale in proportion to perceived heat pain intensity and not temperature intensity during testing.

Determination of the Individualized Test Temperature (ITT): To determine ITT the first temperature stimulus will ramp from baseline (32°C) to 46°C (the 75th percentile heat pain detection threshold for children ages 7-17 years) and held for 5 seconds.[22] The temperature will return to baseline (32°C) for 30 seconds and be repeated three times. If an eVAS of 75/100mm is not consistently reported on all three trials, this paradigm will be repeated at 48ºC. The lowest temperature that consistently evokes an eVAS 75/100mm will be used as the first temperature in all tests.

Offset Analgesia (OA) Test: We will use the same paradigm as our previous study, except for increasing the ITT threshold to 75/100mm.[37] The first temperature (T1) is set to the ITT and held for 5 seconds, followed by a second temperature (T2) 1°Celsius (C) higher for 5 seconds, and then returns to a third temperature (T3) that is equal to T1 for 20 seconds before returning to baseline (32ºC). OA responses are calculated as a percentage of perceived pain reduction following the 1ºC noxious thermal stimulus offset. A larger OA response (i.e., greater pain reduction) reflects a greater ability to actuate pain inhibition.

Control Test: For control tests, T1 and T2 temperatures are identical to those used in the OA paradigm, but T3 is set at the non-noxious baseline temperature (32°C). The control test serves as a physiological discriminative stimulus to examine participants' pain perception in the presence versus absence of a noxious heat stimulus.

Constant Test: For constant tests, the ITT (T1) is applied and held for 30 seconds before returning to baseline (32ºC). The constant test compares the magnitude of habituation and summation occurring during constant and OA tests.

Cardiovascular Endurance Assessment: The Fitkids Treadmill Test (FTT) is a reliable and valid measure of pediatric submaximal cardiovascular endurance.[16; 17] Time to exhaustion (TTE) on the FTT provides an objective, norm-referenced marker of cardiovascular endurance in youth ages 6-18 years and is defined as the total time completed on the test, excluding the warm-up and cool-down phases. Our recent study demonstrated that youth with chronic pain demonstrate impaired cardiovascular endurance compared to age and sex matched peers at baseline and improves significantly after IIPT.[36] The FTT is completed at PPRC admission and discharge as per standard of care for participants who can safely ambulate on a treadmill.

Biopsychosocial Characteristics: A battery of psychosocial and clinical questionnaires are administered as part of routine clinical care at the Mayo Family PPRC and stored in an IRB approved data registry for which Dr. Shulman and Dr. Sethna are co-investigators (P-0015943). Data for responses to these questionnaires will be shared for the current protocol to reduce participant burden. These measures include reliable and valid pediatric questionnaires of physical and emotional functioning including: Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Anxiety short form 8a ,[42] PROMIS Depressive Symptoms short form 8a,[42] PROMIS Pediatric Pain Interference short form 8a,[42] Central Sensitization Inventory,[27; 28] Functional Disability Inventory.[21; 43] Participant characteristics at IIPT admission including, age, sex, diagnosis, pain intensity ratings, time since symptom onset, and medications will also be included to evaluate similarities and differences among OA responders and non-responders for Aim 3 based on prior research.[23; 25; 33; 39]

ELIGIBILITY:
Inclusion Criteria:]

i) age 10-17 years

ii) first test completed within 5 days of admission

iii) established diagnosis of primary or secondary chronic pain

iv) report of constant moderate pain (≥ 5/10 on a numeric rating scale of 0-10 points) for at least 3 months duration

v) stable use of medications for at least one week prior to the study visit.

Exclusion Criteria:

i) presence of allodynia in either upper extremity

ii) a history of central nervous system, heart, kidney, liver and respiratory system diseases, and psychiatric disorders (e.g., bipolar, conversion, psychosis)

iii) reported consumption of alcohol, cannabis or tobacco products

iv) unable to read English or follow testing instructions

v) intolerant to the thermal test stimulus, or vi) no pain reported at maximum stimulus (48ºC).

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Youth with all types of chronic pain syndromes (including but not limited to: headaches, abdominal pain, complex regional pain syndrome, amplified pain syndrome) admitted to the Mayo Family Pediatric Pain Rehabilitation Center for intensive interdisciplinary pain treatment.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Change in Offset Analgesia | through study completion, an average of 4-6 weeks
  Percent reduction in pain following the small, 1º C stimulus offset.

SECONDARY OUTCOMES:
Change in Control Test Response | through study completion, an average of 4-6 weeks
  Percent reduction in pain following a large stimulus offset to a non-noxious temperature.
Change in Constant Test Response | through study completion, an average of 4-6 weeks
  Pain response (area under the curve) during a 30 second constant, moderate heat pain stimulus.
Change in Cardiovascular Endurance | through study completion, an average of 4-6 weeks
  Total time to exhaustion (minutes) on the Fitkids Treadmill Test.

OTHER OUTCOMES:
Change in Anxiety | through study completion, an average of 4-6 weeks
  PROMIS Pediatric Anxiety short form 8a T-score, range 0-100, higher scores = higher anxiety
Change in Depressive Symptoms | through study completion, an average of 4-6 weeks
  PROMIS Depressive Symptoms short form 8a T-score, range = 0-100; higher scores = more depressive symptoms
Change in Pain Interference | through study completion, an average of 4-6 weeks
  PROMIS Pain Interference short form 8a T score; range 0-100; higher scores = higher pain interference
Change in Central Sensitization | through study completion, an average of 4-6 weeks
  Central Sensitization Inventory Total Score (0-100), higher scores = more central sensitization

CONTACTS AND LOCATIONS:
Overall Officials: Julie M Shulman, PT, PhD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hospital at Waltham, Waltham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shulman J, Zurakowski D, Keysor J, Jervis K, Sethna NF. Offset analgesia identifies impaired endogenous pain modulation in pediatric chronic pain disorders. Pain. 2020 Dec;161(12):2852-2859. doi: 10.1097/j.pain.0000000000001984. PMID 32658151
- [Background] Kotte EM, de Groot JF, Bongers BC, Winkler AM, Takken T. Fitkids Treadmill Test: Age- and Sex-Related Normative Values in Dutch Children and Adolescents. Phys Ther. 2016 Nov;96(11):1764-1772. doi: 10.2522/ptj.20150399. Epub 2016 May 19. PMID 27197825
- [Background] Grill JD, Coghill RC. Transient analgesia evoked by noxious stimulus offset. J Neurophysiol. 2002 Apr;87(4):2205-8. doi: 10.1152/jn.00730.2001. PMID 11929939
- [Background] King S, Chambers CT, Huguet A, MacNevin RC, McGrath PJ, Parker L, MacDonald AJ. The epidemiology of chronic pain in children and adolescents revisited: a systematic review. Pain. 2011 Dec;152(12):2729-2738. doi: 10.1016/j.pain.2011.07.016. PMID 22078064
- [Background] Hermans L, Calders P, Van Oosterwijck J, Verschelde E, Bertel E, Meeus M. An Overview of Offset Analgesia and the Comparison with Conditioned Pain Modulation: A Systematic Literature Review. Pain Physician. 2016 Jul;19(6):307-26. PMID 27454261